CLINICAL TRIAL: NCT04627194
Title: Epidemiological and Clinical Characteristics of COVID-19 Patients in Kazakhstan in Early 2020: a Retrospective, Observational Cohort Study
Brief Title: Characteristics of COVID-19 Patients in Kazakhstan in Early 2020
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Semey State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 76.29.31_48.04.06-01
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Pneumonia, Viral
MeSH Terms: conditions — COVID-19; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Mild and asymptomatic COVID-19 patients: Symptomatic patients meeting the World Health Organization (WHO) case definition for COVID-19 without evidence of viral pneumonia or hypoxia, who have a laboratory-confirmed SARS-CoV-2 infection, or asymptomatic patients with a laboratory-confirmed SARS-CoV-2 infection at the time of hospitalization.
- Moderate severity COVID-19 patients: Symptomatic patients with a laboratory-confirmed SARS-CoV-2 infection, meeting the WHO case definition for moderate COVID-19 disease severity [including clinical signs of pneumonia e.g. fever, cough, dyspnoea, fast breathing, but no signs of severe pneumonia] at the time of hospitalization.
- Severe-to-critical COVID-19 patients: Symptomatic patients with a laboratory-confirmed SARS-CoV-2 infection, meeting the WHO case definition(s) for severe COVID-19 disease presentation [including clinical signs of pneumonia e.g. fever, cough, dyspnoea, fast breathing, and one of the following: respiratory rate > 30 breaths/min; severe respiratory distress; or oxygen saturation (SpO2) < 90% on room air] or for critical COVID-19 disease presentation [including acute respiratory distress syndrome (ARDS), sepsis, septic shock or other complications such as acute pulmonary embolism, acute coronary syndrome, acute stroke and delirium] at the time of hospitalization.
- COVID-19 survivors: Patients diagnosed with a laboratory-confirmed COVID-19, who survived.
- COVID-19 non-survivors: Patients diagnosed with a laboratory-confirmed COVID-19, who did not survive.

SUMMARY:
The aim of this study is to assess the epidemiological and clinical features of patients diagnosed with COVID-19 in Kazakhstan at the onset of the pandemic.

DETAILED DESCRIPTION:
There is a paucity of data available on the epidemiological and clinical characteristics of coronavirus disease 2019 (COVID-19) in Kazakhstan. While a global effort in search for effective treatments and vaccines against COVID-19 is in effect, it is important that high quality and up-to-date information be available from a broad variety of populations on the dynamics of infection. This is especially important in regions where, due to resource shortage, epidemiologic surveillance may have gaps. To address the current gaps, medical records will be obtained for patients with confirmed COVID-19 during the first months of the pandemic (February-April 2020). The epidemiologic and clinical features including the demographics, clinical manifestation, laboratory parameters, radiologic assessments and clinical outcomes will be analyzed. The results of this study will facilitate the clinical management of COVID-19 patients in Kazakhstan and ultimately inform the ongoing efforts to curb the spread of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in the region.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmation of SARS-CoV-2 infection by polymerase chain reaction.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical records will be obtained for all subjects, who presented with COVID-19-like symptoms or had a suspected exposure to SARS-CoV-2 between Feb 20 and April 30, 2020 as reported to the Republican Centre for Health Development by regional hospitals. Only those patients who had a positive SARS-CoV-2 PCR test result will be included in the analysis of primary and secondary outcome measures.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and demographic predictors of disease severity among hospitalized COVID-19 patients. | approximately 70 days
  Risk factors associated with disease severity and their odds ratios (ORs) will be assessed by the univariable and multivariable logistic regression models.
Clinical and demographic predictors of mortality among hospitalized COVID-19 patients. | approximately 70 days
  Risk factors associated with death and their odds ratios (ORs) will be assessed by the univariable and multivariable logistic regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Yersin Zhunussov, MD, D.M.S., Study Chair — Semey State Medical University; Raifa Ivanova, MD, D.M.S., Study Director — Semey State Medical University; Maiya Goremykina, M.D, C.M.S, Principal Investigator — Semey State Medical University; Sergey Yegorov, Ph.D., Principal Investigator — Nazarbayev University, School of Sciences and Humanities
Locations (1):
- Semey Medical University, Semey, East Kazakhstan, Kazakhstan

IPD SHARING:
Plan to Share IPD: No